CLINICAL TRIAL: NCT06786767
Title: A Prospective Non-interventional Real-world Study Assessing the Effectiveness of Extrafine BDP/FF/G (Beclometasone Dipropionate/Formoterol Fumarate/Glycopyrronium) 172/5/9 mcg, (Pressurised Inhalation, Solution) Single Inhaler Triple Therapy (SITT) on Symptom Scores in Asthma Patients After 6 Months Treatment
Brief Title: Fixed Triple Inhaled Combination in Asthmatic Patients in a Real-life Setting
Acronym: STRENGTH
Status: Active, not recruiting | Type: Observational
Sponsor: Chiesi Bulgaria (Industry)
Responsible Party: Sponsor
Other Study IDs: BG.MED.TRIHS.24.07.01; НИП-0008/4.11.2024 (Other: Ministry of Health, Bulgarian Drug Agency); CT-0727/06.11.2024 (Other: Ministry of Health; Ethics committee for Clinical Trials)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Asthma; Asthma Patients; Asthma Bronchiale
Keywords: Asthma therapy; Fixed triple inhalation treatment; Trimbow
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asthmatic patients switched to Trimbow (BDP/FF/G 172/5/9 μg): Asthmatic patients switched to BDP/FF/G 172/5/9 μg before study enrollment or at the day of enrollment due to uncontrolled asthma (a) patients who experienced one or more asthma exacerbation in the previous year and uncontrolled despite the use of b1) LABA and high dose ICS or b2) LABA and high-dose ICS + LAMA multi-inhaler triple therapy.
  Interventions: Drug: BDP/FF/G (Beclomethasone diprprionate, formoterol fumarate, glycopyrronium bromide) 172/5/9 μg

INTERVENTIONS:
Drug: BDP/FF/G (Beclomethasone diprprionate, formoterol fumarate, glycopyrronium bromide) 172/5/9 μg — As this is a non-interventional study, it is accordance with routing clinical practice. The assignment of patients to Trimbow 172/5/9 mcg should be made independently from the study.

SUMMARY:
The mainstay of asthma treatment are ICSs, mostly and usually combined with LABA. In the past decade LAMA had been accepted as an add-on treatment for patients on GINA treatment Steps 4 and 5. Recently, RCTs proved the efficacy and safety of fixed triple combinations of moderate and high dose of ICS and LABA, LAMA in a very selected asthmatic population, resulting in the market authorization of these products. However, there is a lack of evidence on the real-world effectiveness of these therapies, especially with regards to improvement in symptom scores and quality of life.

DETAILED DESCRIPTION:
Study design: multicenter, national, non-interventional, prospective study evaluating the effectiveness of Trimbow 172/5/9 μg pMDI on symptom scores in 6 months after switch from previous LABA-high dose ICS or LABA-high dose ICS + LAMA containing treatment in asthmatic patients.

Dosage regimen and administration Name of the product: Trimbow 172/5/9 micrograms pressurised inhalation, solution. Each delivered dose (the dose leaving the mouthpiece) contains 172 μg of beclometasone dipropionate, 5 μg of formoterol fumarate dihydrate and 9 μg of glycopyrronium (as 11 μg glycopyrronium bromide). Each metered dose (the dose leaving the valve) contains 200 μg of beclometasone dipropionate, 6 μg of formoterol fumarate dihydrate and 10 μg of glycopyrronium (as 12.5 μg glycopyrronium bromide). The recommended dose is two inhalations twice daily. The maximum dose is two inhalations twice daily.

1. Aim of the study (research objective)

   Primary objective:

   The main objective is to assess the effectiveness of BDP/FF/G 172/5/9 μg fixed triple combination in a real-world setting, with regards to improvements in symptom scores (ACT - Asthma Control Test).

   Primary outcome measures:
   * Change (improvement) of ACT score, during the 6 months of treatment (Visit 3), compared to the score at baseline.
   * The percentage of patients achieving an improvement in ACT score of 3 points (MCID, minimum clinically important difference) or more, after the 6-month treatment (Visit 3) compared to baseline.

   Secondary objectives:

   Secondary objectives are the assessments of improvement in lung function, adherence to treatment, and health-related quality of life.
2. Test sample and method, recruitment principle No patient recruitment will be performed. Eligible patients will be enrolled during the participating physicians' regular asthma patient management and patients' written informed consent. Patient inclusion will take place among patients having severe asthma at outpatient clinics (the chosen study sites are attached as annexes to the study protocol), strictly at the time of the patients' visit. The planned number of patients is up to 300.
3. Structure of the study In accordance with the requirements of non-interventional studies, the assignment of patients to Trimbow 172/5/9 μg pMDI therapy should be made independently of the study. Patient enrolment can take place after the patient has been fully informed about the purpose of the study and all its details, and the patient has read and signed the patient informed consent form, including any questions they may have. Once this has taken place, the data that would have been generated anyway during the outpatient examination of the patient in accordance with daily practice can be recorded. This is considered the first visit of the study (Visit 1). During this visit, the patient's main demographic data, information on comorbidities and concomitant medications, smoking history, previous and current asthma therapies, asthma specific assessment (including ACT), exacerbation history, post-dose lung function values, maintenance and reliever inhaled therapies (former and new) baseline quality of life based on the asthma quality of life (EQ-5D-5L) questionnaire, and adherence to therapy based on Test of Adherence to Inhalers (TAI-12) questionnaire are recorded (data to be recorded in e-CRF). Patients will then attend two additional visits - Visit 2 - 1 month (30 ± 5 days) and Visit 3 - 6 months ± 10 days after enrolment as per routine clinical practice. During these visits, data will be collected, according to routine clinical practice. If the patient's maintenance therapy changes during the study as decided by the treating physician, and the patient is no longer receiving Trimbow 172/5/9 μg pMDI, the patient will be automatically excluded from this NIS. The therapy modification and its exact date must be recorded in the eCRF (electronic Case Report Form) of the next visit. If the change in therapy is related to a suspected adverse reaction, it should be reported separately in the eCRF platform in accordance with the respective section of the protocol.

   This NIS is open to all eligible patients according to the inclusion and exclusion criteria. Permitted concomitant treatments: allowed all medications according to local clinical practice (any non-inhalation therapy for asthma or other diseases) and reliever (short-acting bronchodilators) inhaled therapies for asthma.
4. Start and duration of the study The enrolment of the patients can start only after the approval of the Bulgarian Drug Agency and Ethics Committee for Clinical Trials. The study is planned to start at the end of January 2025. Each site will have 3 months to enroll patients. Following the completion of patient enrolment, each patient will be followed up for 6 months. After the visit of the last patient, sites will have one month to collect all missing data/correct any data flagged as erroneous during monitoring. The last patient last visit is expected to take place in October/November 2025, and the study is planned to be concluded in March/April 2026.
5. Study plan A total of 3 visits will be performed for the assessment of the primary and secondary endpoints during the study. Patients may be enrolled in the study and their data may be recorded, only if this data is recorded in accordance with standard medical practice.

   * Visit 1: time of enrolment - a normal visit, according to routine clinical practice. Informed consent and baseline patient characteristics will be collected.
   * Visit 2: 1 month after enrolment (30 days ± 5 days after Visit 1)
   * Visit 3: 6 months after enrolment (± 10 days).

ELIGIBILITY:
Inclusion Criteria:

1. Physician-confirmed clinical diagnosis of asthma according to GINA guidelines and treated for at least 3 years before inclusion
2. Patients ≥ 18 years of age in ambulatory care
3. Patients who are eligible for the use of Trimbow 172/5/9 μg pMDI according to the SmPC

   1. patients who experienced one or more asthma exacerbation in the previous year AND
   2. patients not adequately controlled according to the physician's clinical assessment despite the use of b1) LABA and high dose ICS OR b2) LABA and high-dose ICS + LAMA multi-inhaler triple therapy. FEV1<80% at baseline. (spirometry performed at the visit 1 independently of the study or up to 30 days before the enrolment or within 3 days after Visit 1 is acceptable).

5. Inhaled asthma therapy was changed to Trimbow 172/5/9 μg pMDI no more than 2 weeks prior to OR on the day of study inclusion 6. Patient provided written, informed consent to study participation

Exclusion Criteria:

1. Participation in any clinical trial within 30 days prior to enrolment
2. Patients hospitalized due to an exacerbation of their asthma within the last 4 weeks prior to enrolment.
3. Diagnosis of COPD.
4. Tuberculosis (active or anamnestic)
5. Actual or previous use of biologics for asthma treatment in the past 12 months
6. All exclusion criteria listed in Trimbow 172/5/9 μg pMDI SmPC
7. Hypersensitivity to the active substances or to any of the excipients listed in the SmPC
8. Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient inclusion will take place among patients having severe asthma at outpatient clinics in the selected and approved sites.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test | 6 months
  Change (improvement) of Asthma Control Test score, during the 6 months of treatment (Visit 3), compared to the score at baseline. A maximum score of 25 points indicates complete asthma control, while a score less than 16 indicates very poorly controlled asthma.
Asthma Control Test - 2 | 6 months
  The percentage of patients achieving an improvement in Asthma Control Test score of 3 points (MCID, minimum clinically important difference) or more, after the 6-month treatment (Visit 3) compared to baseline. A maximum score of 25 points indicates complete asthma control, while a score less than 16 indicates very poorly controlled asthma.

SECONDARY OUTCOMES:
Asthma Control Test change | 6 months
  The percentage of patients achieving an improvement according to asthma control levels (uncontrolled= ACT ≤15; partially controlled= 15<ACT<20; controlled 20≤ACT).
HRQoL | 6 months
  Change in Health-related QoL was assessed by measuring the 5-level EuroQoL 5-dimension component (EQ-5D-5L) index score at Visit 3 (6 months), compared to the baseline visit 1 (Week 0), regarding the assessment of the impact of Asthma on the patient's quality of life. (levels 1 to 5; 1 = indication no problem; 5 = indicating unable to/extreme problems).
Test of Adherence to Inhalers (TAI-12) | 6 months
  Change in Test of Adherence to Inhalers (TAI-12) score at Visit 3 (6 months) compared to baseline visit (Visit 1, week 0) regarding adherence to treatment with use of the Trimbow 172/5/9 μg pMDI (50 points = good adherence; 46 to 49 points = intermediate adherence; < 45 points = poor adherence).
Lung function | 6 months
  Change in spirometry parameters: FEV1, FVC, FEV1/FVC, at Visit 3 (6 months), compared to the baseline Visit 1 (Week 0), with use of the Trimbow 172/5/9 μg pMDI.

CONTACTS AND LOCATIONS:
Overall Officials: Yavor Y. Ivanov, Asso.Prof., Study Chair — Group practice for specialized medical care - Asthma Center Pleven; Neli L. Rodopska, Pharm.M.Sc, Study Director — Chiesi Bulgaria
Locations (14):
- Bulgaria (14):
  - AIPSMCPP Dr. Elina Smilkova, Blagoevgrad
  - Medical Center Viva Phenix, Dobrich
  - Medical Center Hipocrat, Gabrovo
  - ASIMPIDPP Dr. Veselin Kalfov, Haskovo
  - Medical Center Denitza, Montana
  - IPASMC Dr. Kostadinka Sotirova, Pazardzhik
  - Group practice for specialized medical care - Asthma Center Pleven, Pleven
  - AIPSACA Dr. Talyat Cholak, Razgrad
  - AIPSMC Dr. Svetlan Mihaylov, Stara Zagora
  - Medical Center Third Policlinic, Stara Zagora
  - MHAT Svoge, Svoge
  - AIPSMCPP Dr. Nikolay Lichev V. Tarnovo, Veliko Tarnovo
  - Medical Center St. Ivan Rilski, Vidin
  - AIPSMCPP Dr. Bilyana Ivanova, Vratsa

IPD SHARING:
Plan to Share IPD: No
IDP is sole property of the sponsor and will only be eligible upon reasonable request.